CLINICAL TRIAL: NCT00369954
Title: A Phase II Trial of Intravenous Gemcitabine (NSC #613327) and Intraperitoneal Carboplatin (NSC # 241240) in the Treatment of Patients With Platinum-Sensitive Epithelial Ovarian, Primary Peritoneal, or Fallopian Tube Carcinoma With Non-Measurable Disease
Brief Title: Gemcitabine and Carboplatin in Treating Patients With Persistent or Recurrent Ovarian Epithelial Cancer, Primary Peritoneal Cancer, or Fallopian Tube Cancer That Responded to Previous Cisplatin or Carboplatin
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial was never activated
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Philip J. DiSaia, Gynecologic Oncology Group
Organization: GOG Foundation (Network)
Purpose: Treatment
Other Study IDs: CDR0000496764; GOG-0102H
Record Dates: First submitted 2006-08-29; First posted 2006-08-30 (Estimated); Last update posted 2013-06-10 (Estimated); Status verified 2007-10

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Peritoneal Cavity Cancer
Keywords: recurrent ovarian epithelial cancer; fallopian tube cancer; peritoneal cavity cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Carboplatin; Gemcitabine

INTERVENTIONS:
Drug: carboplatin
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) and giving them in different ways may kill more tumor cells.

PURPOSE: This phase II trial is studying the side effects and how well giving gemcitabine together with carboplatin works in treating patients with persistent or recurrent ovarian epithelial cancer, primary peritoneal cancer, or fallopian tube cancer that responded to previous cisplatin or carboplatin.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the progression-free survival of patients with persistent or recurrent platinum-sensitive ovarian epithelial, fallopian tube, or primary peritoneal cancer treated with gemcitabine hydrochloride and intraperitoneal carboplatin.
* Evaluate the systemic and regional toxicity of this regimen in these patients.

Secondary

* Determine the overall survival of patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive gemcitabine hydrochloride IV over 30 minutes followed by intraperitoneal carboplatin on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 3 years.

PROJECTED ACCRUAL: A total of 100 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed ovarian epithelial cancer, primary peritoneal cancer, or fallopian tube cancer

  * Persistent or recurrent disease
* Nonmeasurable disease
* Platinum-sensitive disease

  * Must have attained a clinically defined complete response after prior platinum- (cisplatin or carboplatin) and taxane-based combination chemotherapy regimen

    * Patients with partial response or disease progression after first-line therapy are not eligible
    * No disease recurrence within 6 months after completion of first-line platinum-taxane therapy
* Must have undergone laparoscopy or laparotomy for either of the following:

  * Second-look surgery after a complete response to first-line therapy

    * No negative second-look surgery
  * Secondary cytoreductive surgery for recurrent disease ≥ 6 months after completion of first-line chemotherapy
* No greater than 1 cm residual disease at the completion of laparoscopy or laparotomy AND no diffuse carcinomatosis
* Disease must be confined to the peritoneal cavity

  * Retroperitoneal disease ≤ 1 cm at the completion of prior surgery allowed
* Not a candidate for a higher priority GOG protocol
* No tumors of low malignant potential

PATIENT CHARACTERISTICS:

* GOG performance status 0-2
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN
* SGOT ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN
* Neuropathy (sensory and motor) ≤ grade 1
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active infection requiring antibiotics
* No other invasive malignancies within the past 5 years except nonmelanoma skin cancer
* No extensive intra-abdominal adhesions

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from prior surgery or chemotherapy
* No prior intraperitoneal therapy
* No prior gemcitabine hydrochloride
* No more than 1 prior regimen (including consolidation chemotherapy) for ovarian epithelial cancer, primary peritoneal cancer, or fallopian tube cancer
* No radiotherapy to > 25% of marrow-bearing areas
* No prior abdominal-pelvic radiotherapy
* No prior cancer treatment that would preclude study therapy
* No other prior therapy directed at the malignant tumor, including biological agents (unless this was part of front-line therapy), immunologic agents, vaccines, second-line chemotherapy, or hormonal therapy

  * Concurrent hormone replacement therapy allowed
* No concurrent amifostine or other protective reagents

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-04

PRIMARY OUTCOMES:
Relative risk of progression-free survival
Frequency and severity of observed adverse effects by CTCAE version 3.0

SECONDARY OUTCOMES:
Relative risk of survival

CONTACTS AND LOCATIONS:
Overall Officials: Noelle G. Cloven, MD, Study Chair — Methodist Estabrook Cancer Center